CLINICAL TRIAL: NCT00755053
Title: An Investigator-blinded, Active-controlled Phase 3 Study to Prove the Non-inferior Efficacy of a Clotrimazole Ovule (500 mg) Versus a Clotrimazole Vaginal Tablet (500 mg) in Vaginal Candidiasis
Brief Title: Comparative Efficacy of Ovule vs Tablet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13071; 2008-000718-63 (EudraCT Number)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-07

CONDITIONS: Clotrimazole; Ovulen; Vulvovaginal Candidiasis
Keywords: Clotrimazole; Ovule; Tablet; Vulvovaginal candidiasis; Non-inferiority
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clotrimazole tablet (Canesten, BAY-B5097) (Active Comparator): Single intravaginal dose of 500 mg clotrimazole tablet at Visit 1 (Day 0).
  Interventions: Drug: Clotrimazole, vaginal tablet
- Clotrimazole ovule (Canesten, BAY-B5097) (Experimental): Single intravaginal dose of 500 mg clotrimazole ovule at Visit 1 (Day 0).
  Interventions: Drug: Clotrimazole, vaginal ovule

INTERVENTIONS:
Drug: Clotrimazole, vaginal ovule — Single intravaginal dose of 500 mg clotrimazole ovule at Visit 1 (Day 0).
  Arms: Clotrimazole ovule (Canesten, BAY-B5097)
Drug: Clotrimazole, vaginal tablet — Single intravaginal dose of 500 mg clotrimazole tablet at Visit 1 (Day 0).
  Arms: Clotrimazole tablet (Canesten, BAY-B5097)

SUMMARY:
The study is focused to prove that the efficacy of a new Canesten formulation (ovule) is not inferior to the old Canesten formulation (tablet)

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant females aged at least 14 years in Germany or at least 16 years in Russia and not older than 50 years.
* Subjects presenting a symptomatic vulvovaginal yeast infection confirmed by microscopic evaluation (wet mount preparation).
* Subjects must be cooperative, able to understand the requirements of the trial participation, and willing to participate in the trial. For adolescents the informed consent has to be provided to a legal representative in addition.
* Subjects of childbearing potential must use an acceptable method of contraception. Hormonal or oral contraceptive drugs, intra-uterine devices (IUD) and abstinence are considered acceptable methods of contraception.
* Negative saline smear for Trichomonas vaginalis

Exclusion Criteria:

* Subjects with known hypersensitivity to imidazoles or triazoles and their analogues.
* Subjects presenting a protozoan infection as confirmed by microscopic investigation.
* Pregnant, breast feeding or lactating subjects.
* Subjects with suspected bacterial vaginal infection.
* Subjects with abdominal pain, fever, or foul smelling vaginal discharge.
* Subjects who had a vaginal infection, or who had used an intravaginal or systemic antimycotic treatment within 60 days prior to visit 1.
* Subjects using or wishing to use intra-vaginal or systemic anti-infectives or systemic antifungal therapy during the trial.
* Subjects wishing to use contraceptive foams, creams, jellies, sponges, therapeutic ointments, condoms, diaphragms, and OTC vaginal products during treatment and 3 days thereafter (i.e. until day 4).
* Subjects unable to refrain from the use of vaginal tampons during treatment and for 3 days thereafter (i.e. until day 4).
* Subjects unable to refrain from the use of feminine hygiene products (e.g. douches, feminine deodorant products) for 2 weeks (i.e. from visit 1 until visit 2).
* Subjects suffering from chronic/recurrent vulvovaginal mycosis, defined as 4 or more mycologically proven symptomatic episodes during the last 12 months.
* Subjects suffering from diseases (e.g. diabetes, decreased cellular immunity) or being treated with drugs (e.g. immunosuppressants, corticosteroids, anti-infectives) which may predispose them to mycological infections.
* Subjects who received another investigational drug within 30 days before visit 1.
* Unwillingness to refrain from sexual activity during 3 days thereafter.
* Actual menstruation at visit 1 or expected menstruation within 4 days after visit 1.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 466 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects With Overall Response at Visit 2 (Day 10 to 14) | 10-14 days after treatment (=visit 2)

SECONDARY OUTCOMES:
Percentage of Subjects With Overall Response at Visit 3 (Week 6 to 8) | 6-8 weeks after treatment (=visit 3)
Percentage of Subjects With Clinical Cure at Visit 2 (Day 10 to 14) | 10-14 days after treatment (=visit 2)
Percentage of Subjects With Clinical Cure at Visit 3 (Week 6 to 8) | 6-8 weeks after treatment (=visit 3)
Percentage of Subjects With Mycological Cure at Visit 2 (Day 10 to 14) | 10-14 days after treatment (=visit 2)
Percentage of Subjects With Mycological Cure at Visit 3 (Week 6 to 8) | 6-8 weeks after treatment (=visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Germany (10):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - München, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Wiesbaden, Hesse
  - Hanover, Lower Saxony
  - Osnabrück, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Krefeld, North Rhine-Westphalia
- Moscow, Russia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu